CLINICAL TRIAL: NCT02548767
Title: Adverse Metabolic Effects of Dietary Sugar: Ad Libitum vs Energy-balanced Diets
Brief Title: Adverse Metabolic Effects of Dietary Sugar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Touro University, California (Other); University of Southern California (Other); USDA, Western Human Nutrition Research Center (U.S. Federal Agency); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 499106; 1R01HL121324 (NIH)
Record Dates: First submitted 2015-05-26; First posted 2015-09-14 (Estimated); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Chronic Disease of Cardiovascular System; Type 2 Diabetes; Obesity
Keywords: High fructose corn syrup; Sugar
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity | interventions — High Fructose Corn Syrup; Sugars; Aspartame

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- HFCS-EB (Experimental): Consume 3 servings/day of high fructose corn syrup (HFCS)-sweetened beverage along with the provided energy-balanced diet. The 3 HFCS-sweetened beverages will contain 25% of energy requirement and the remainder of the provided diet will contain 75% of energy requirement. All and only the provided beverage and diet will be consumed for eight weeks.
  Interventions: Other: high fructose corn syrup; Other: Energy-balanced diet
- Asp-EB (Placebo Comparator): Consume 3 servings/day of aspartame-sweetened beverage along with the provided energy-balanced diet. The 3 aspartame-sweetened beverages will contain 0% of energy requirement and the remainder of the provided diet will contain 100% of energy requirement. All and only the provided beverage and diet will be consumed for eight weeks.
  Interventions: Other: aspartame; Other: Energy-balanced diet
- HFCS-AL (Experimental): Consume 3 servings/day of high fructose corn syrup (HFCS)-sweetened beverage along with the provided ad libitum diet. The 3 HFCS-sweetened beverages will contain 25% of energy requirement and the remainder of the provided diet will contain approximately 125% of energy requirement. All the provided beverage will be consumed for eight weeks. Only the provided beverage and diet will be consumed for eight weeks. The provided diet will be consumed ad libitum and the uneaten portions will be returned to study staff.
  Interventions: Other: high fructose corn syrup; Other: Ad libitum diet
- Asp-AL (Placebo Comparator): Consume 3 servings/day of aspartame-sweetened beverage along with the provided ad libitum diet. The 3 aspartame-sweetened beverages will contain 0% of energy requirement and the remainder of the provided diet will contain approximately 125% of energy requirement. All the provided beverage will be consumed for eight weeks. Only the provided beverage and diet will be consumed for eight weeks. The provided diet will be consumed ad libitum and the uneaten portions will be returned to study staff.
  Interventions: Other: aspartame; Other: Ad libitum diet

INTERVENTIONS:
Other: high fructose corn syrup — High fructose corn syrup provided as 15% HFCS/85% water (weight/weight) fruit-flavored beverage
  Other Names: sugar, HFCS, high fructose corn syrup-55, HFCS-55
  Arms: HFCS-AL; HFCS-EB
Other: aspartame — Aspartame provided as 0.04% aspartame/99.96% water (weight/weight), fruit-flavored beverage
  Other Names: non-caloric sweetener
  Arms: Asp-AL; Asp-EB
Other: Energy-balanced diet — Provided in quantities that equal energy requirement. Formulated such that the overall macronutrient intake; including beverage; equal 45%/5% energy requirement at complex/simple carbohydrate, 35% energy requirement as fat, 15% energy requirement as protein.
  Other Names: Weight-maintaining diet
  Arms: Asp-EB; HFCS-EB
Other: Ad libitum diet — Provided in quantities that exceed energy requirement by approximately 25%. Formulated such that the overall macronutrient intake; including beverage; equals approximately 45%/5% energy requirement at complex/simple carbohydrate, 35% energy requirement as fat, 15% energy requirement as protein.
  Other Names: Positive-energy diet
  Arms: Asp-AL; HFCS-AL

SUMMARY:
It is not known whether consumption of excessive amounts of sugar can increase risk factors for cardiovascular disease or diabetes in the absence of increased food (caloric) intake and weight gain, nor whether the negative effects of sugar consumption are made worse when accompanied by weight gain. This study will investigate the effects of excess sugar when consumed with an energy-balanced diet that prevents weight gain, and the effects of excess sugar when consumed with a diet that can cause weight gain. The results will determine whether excess sugar consumption and excess caloric intake that lead to weight gain have independent and additive effects on risk factors for cardiovascular disease or diabetes, and will have the potential to influence dietary guidelines and public health policy.

DETAILED DESCRIPTION:
Recent studies have demonstrated that consuming high fructose corn syrup (HFCS)- or sucrose-sweetened beverages increased lipid/lipoprotein risk factors for cardiovascular disease (CVD) in healthy adults compared with iso-caloric amounts of glucose or low-fat milk. The longest of these studies, which utilized a 6-month intervention, also showed increased liver and muscle TG and increased visceral adipose deposition. Neither of these studies found differences in weight gain between subjects consuming HFCS/sucrose beverages compared with control beverages. These results suggest that it is not just excess calories and weight gain that mediate the effects of dietary sugar/fructose on the development of metabolic disease; rather, dietary sugar per se is also a contributor. However, it is not known whether consumption of excessive amounts of sugar can increase risk factors for metabolic disease in the absence of positive energy balance and weight gain, nor whether the adverse effects of sugar consumption are exacerbated by weight gain. This study will compare the contribution of sugar with the contribution of energy level to the increases in risk factors for metabolic disease induced by consumption of HFCS-sweetened beverages under energy-balanced or ad libitum conditions. The investigators will measure risk factors and processes associated with metabolic disease in 4 groups of young, healthy adults who will consume 1) 0%, 2) or 25% of energy requirement as HFCS-sweetened beverages for 8 weeks with an energy-balanced diet for 6 weeks; 3) 0%, or 4) 25% of energy requirement as HFCS-sweetened beverages for 8 weeks with an ad libitum diet for 6 weeks. All diets, formulated to achieve a comparable macronutrient intake (55% energy as carbohydrate, 35% fat, 15% protein) among all 4 experimental groups, will be provided to the subjects throughout the entire study. The investigators hypothesize that under energy balanced (EB) condition that prevent body weight gain, consumption of HFCS-sweetened beverages will result in adverse metabolic effects compared with aspartame-sweetened beverages. Consumption of HFCS-sweetened beverages with the ad libitum (AL) diet will result in increased energy intake and body weight gain compared with aspartame-sweetened beverages, and will also result in adverse metabolic effects that are more marked than with consumption of HFCS-sweetened beverages with the energy-balanced diet. These results will demonstrate that consumption of HFCS-sweetened beverages increases risk for metabolic disease both directly, via the adverse effects of fructose on lipid and carbohydrate metabolism, and indirectly, via the effects of HFCS-sweetened beverages to promote excess energy intake and body weight gain. These findings will have the potential to influence dietary guidelines and public health policy.

ELIGIBILITY:
Inclusion Criteria:

* BMI 22-28 kg/m2
* Self-reported stable body weight during the prior six months

Exclusion criteria:

* Fasting glucose >105 mg/dl
* Evidence of liver disorder [AST (Aspartate Aminotransferase) or ALT (Alanine Aminotransferase)] >200% upper limit of normal range)
* Evidence of kidney disorder (>2.0mg/dl creatinine)
* Evidence of thyroid disorder (out of normal range)
* Systolic blood pressure consistently over 140mm Hg (mercury) or diastolic blood pressure over 90mmHg
* Triglycerides > 200mg/dl
* LDL-C > 130mg/dl in combination with Chol:HDL > 4
* Hemoglobin < 8.5 g/dL
* Pregnant or lactating women
* Any other condition that, in the opinion of the investigators, would put the subject at risk
* Current, prior (within 12 months), or anticipated use of any hypolipidemic or anti-diabetic agents.
* Use of thyroid, anti-hypertensive, anti-depressant, weight loss medications or any other medication which, in the opinion of the investigator, may confound study results
* Use of tobacco
* Strenuous exerciser (>3.5 hours/week at a level more vigorous than walking)
* Surgery for weight loss
* Diet exclusions: Food allergies, special dietary restrictions, food allergies, routine consumption of less than 3 meals/day, routine ingestion of more than 2 sugar-sweetened beverages or 1 alcoholic beverage/day, unwillingness to consume any food on study menu
* Hydrogen concentration in breath sample following consumption of HFCS-beverage during screening >50ppm
* Veins that are assessed by the CCRC (Clinical Research Center) R.N.s as being unsuitable for long-term infusions and multiple blood draws from a catheter.
* Pre-existing claustrophobia or metal implants that preclude MRI

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2016-02; Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Change of de novo lipogenesis: palmitate tracer-to-tracee ratios by gas chromatography-mass spectrometry. | 22 hours at Baseline and 4-week Intervention
  Blood samples are collected during 26-h isotopic acetate infusion. Blood samples are processed for determination of palmitate tracer-to-tracee ratios by gas chromatography-mass spectrometry.

SECONDARY OUTCOMES:
Change of endogenous glucose production measured by standard dilution techniques | 7 hours at Baseline and 4-week Intervention
  Blood samples are collected during isotopic glucose infusion, and endogenous glucose production (glucose appearance) is measured by standard dilution techniques.
Change of whole body insulin sensitivity | 3 hours at Baseline and 4-week Intervention
  A variable 20% glucose infusion is adjusted to maintain euglycemia during insulin infusion in order to determine insulin-mediated glucose uptake.
Change of liver lipid | Baseline, 4-week Intervention and 8-week intervention
  Quantified from magnetic resonance imaging
Change of fat oxidation | 17 hours at Baseline and 4-week Intervention
  Fat oxidation is calculated from measures of oxygen consumption and carbon dioxide production by indirect calorimetry.
Change of Very low density lipoprotein (VLDL)-triglyceride (TG) kinetics | 22 hours at Baseline and 4-week Intervention
  During overnight fasting VLDL-TG kinetics will be determined using a prime constant infusion of isotopic glycerol. During the meal-feeding protocol, the washout kinetic enrichment of isotopic glycerol in the TG will be used to estimate VLDL-TG with a non-steady modeling approach.

OTHER OUTCOMES:
Change of blood levels of LDL-cholesterol | Baseline and 4-week Intervention
  fasting and postprandial plasma concentrations of TG, cholesterol, low density lipoprotein cholesterol, apolipoprotein B, apolipoprotein C3 are measured
Change of blood levels of non-HDL-cholesterol | Baseline and 4-week Intervention
  fasting and postprandial plasma concentrations of TG, cholesterol, low density lipoprotein cholesterol, apolipoprotein B, apolipoprotein C3 are measured
Change of blood levels of apolipoprotein B | Baseline and 4-week Intervention
  fasting and postprandial plasma concentrations of TG, cholesterol, low density lipoprotein cholesterol, apolipoprotein B, apolipoprotein C3 are measured
Change of blood levels of triglyceride | Baseline and 4-week Intervention
  fasting and postprandial plasma concentrations of TG, cholesterol, low density lipoprotein cholesterol, apolipoprotein B, apolipoprotein C3 are measured
Change of blood levels of apolipoprotein C3 | Baseline and 4-week Intervention
  fasting and postprandial plasma concentrations of TG, cholesterol, low density lipoprotein cholesterol, apolipoprotein B, apolipoprotein C3 are measured
Change of blood levels of uric acid | Baseline and 4-week Intervention
  fasting and postprandial plasma concentrations of uric acid are measured

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Havel, DVM, Ph.D, Principal Investigator — University of California, Davis; Jean-Marc Schwarz, Ph.D., Principal Investigator — Touro University; Kimber L Stanhope, Ph.D., Study Director — University of California, Davis
Locations (3):
- United States (3):
  - University of California, Davis, Davis, California
  - Clinical Research Center, Sacramento, California
  - Touro University California Translational Research Clinic and Student Health Clinic, Vallejo, California

REFERENCES:
- [Background] Stanhope KL, Schwarz JM, Havel PJ. Adverse metabolic effects of dietary fructose: results from the recent epidemiological, clinical, and mechanistic studies. Curr Opin Lipidol. 2013 Jun;24(3):198-206. doi: 10.1097/MOL.0b013e3283613bca. PMID 23594708
- [Background] Cox CL, Stanhope KL, Schwarz JM, Graham JL, Hatcher B, Griffen SC, Bremer AA, Berglund L, McGahan JP, Keim NL, Havel PJ. Consumption of fructose- but not glucose-sweetened beverages for 10 weeks increases circulating concentrations of uric acid, retinol binding protein-4, and gamma-glutamyl transferase activity in overweight/obese humans. Nutr Metab (Lond). 2012 Jul 24;9(1):68. doi: 10.1186/1743-7075-9-68. PMID 22828276
- [Background] Cox CL, Stanhope KL, Schwarz JM, Graham JL, Hatcher B, Griffen SC, Bremer AA, Berglund L, McGahan JP, Havel PJ, Keim NL. Consumption of fructose-sweetened beverages for 10 weeks reduces net fat oxidation and energy expenditure in overweight/obese men and women. Eur J Clin Nutr. 2012 Feb;66(2):201-8. doi: 10.1038/ejcn.2011.159. Epub 2011 Sep 28. PMID 21952692
- [Background] Stanhope KL, Bremer AA, Medici V, Nakajima K, Ito Y, Nakano T, Chen G, Fong TH, Lee V, Menorca RI, Keim NL, Havel PJ. Consumption of fructose and high fructose corn syrup increase postprandial triglycerides, LDL-cholesterol, and apolipoprotein-B in young men and women. J Clin Endocrinol Metab. 2011 Oct;96(10):E1596-605. doi: 10.1210/jc.2011-1251. Epub 2011 Aug 17. PMID 21849529
- [Background] Stanhope KL. Role of fructose-containing sugars in the epidemics of obesity and metabolic syndrome. Annu Rev Med. 2012;63:329-43. doi: 10.1146/annurev-med-042010-113026. Epub 2011 Oct 27. PMID 22034869
- [Background] Stanhope KL, Schwarz JM, Keim NL, Griffen SC, Bremer AA, Graham JL, Hatcher B, Cox CL, Dyachenko A, Zhang W, McGahan JP, Seibert A, Krauss RM, Chiu S, Schaefer EJ, Ai M, Otokozawa S, Nakajima K, Nakano T, Beysen C, Hellerstein MK, Berglund L, Havel PJ. Consuming fructose-sweetened, not glucose-sweetened, beverages increases visceral adiposity and lipids and decreases insulin sensitivity in overweight/obese humans. J Clin Invest. 2009 May;119(5):1322-34. doi: 10.1172/JCI37385. Epub 2009 Apr 20. PMID 19381015
- [Background] Maersk M, Belza A, Stodkilde-Jorgensen H, Ringgaard S, Chabanova E, Thomsen H, Pedersen SB, Astrup A, Richelsen B. Sucrose-sweetened beverages increase fat storage in the liver, muscle, and visceral fat depot: a 6-mo randomized intervention study. Am J Clin Nutr. 2012 Feb;95(2):283-9. doi: 10.3945/ajcn.111.022533. Epub 2011 Dec 28. PMID 22205311
- [Background] Aeberli I, Hochuli M, Gerber PA, Sze L, Murer SB, Tappy L, Spinas GA, Berneis K. Moderate amounts of fructose consumption impair insulin sensitivity in healthy young men: a randomized controlled trial. Diabetes Care. 2013 Jan;36(1):150-6. doi: 10.2337/dc12-0540. Epub 2012 Aug 28. PMID 22933433
- [Background] Schwarz JM, Noworolski SM, Wen MJ, Dyachenko A, Prior JL, Weinberg ME, Herraiz LA, Tai VW, Bergeron N, Bersot TP, Rao MN, Schambelan M, Mulligan K. Effect of a High-Fructose Weight-Maintaining Diet on Lipogenesis and Liver Fat. J Clin Endocrinol Metab. 2015 Jun;100(6):2434-42. doi: 10.1210/jc.2014-3678. Epub 2015 Mar 31. PMID 25825943
- [Derived] Bergwall S, Johansson A, Sonestedt E, Acosta S. High versus low-added sugar consumption for the primary prevention of cardiovascular disease. Cochrane Database Syst Rev. 2022 Jan 5;1(1):CD013320. doi: 10.1002/14651858.CD013320.pub2. PMID 34986271